CLINICAL TRIAL: NCT07008066
Title: Exercise-induced Cardioversion in Persistent Atrial Fibrillation (ExPAF): A Feasibility Pilot Study
Brief Title: Exercise-induced Cardioversion in Persistent Atrial Fibrillation
Acronym: ExPAF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Region Västmanland (Other)
Responsible Party: Principal Investigator, Pär Hedberg, Associate Professor, Senior Consultant, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-01883-01
Record Dates: First submitted 2025-04-23; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Exercise Testing; Persistent Atrial Fibrillation; Electrical Cardioversion; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Standard of Care; Electric Countershock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Patients will undergo a symptom-limited ergometer cycling test under medical supervision. If the atrial fibrillation is not converted to sinus rhythm during the exercise test, the patients will be electrically converted.
  Interventions: Other: Bicycle ergometer excercise
- Control group (Active Comparator): Standard care with planned electrical cardioversion without exercise intervention.
  Interventions: Procedure: Standard care with electrical cardioversion

INTERVENTIONS:
Other: Bicycle ergometer excercise — Patients will undergo a symptom-limited ergometer cycling test under medical supervision. If the atrial fibrillation is not converted to sinus rhythm during the exercise test, the patients will be electrically converted.
  Arms: Exercise group
Procedure: Standard care with electrical cardioversion — Standard care with planned electrical cardioversion without exercise intervention.
  Arms: Control group

SUMMARY:
This study aims to to evaluate the feasibility of conducting a larger randomized controlled trial (RCT) to assess whether an exercise stress test on an ergometer bicycle could induce sinus rhythm in patients with persistent AF scheduled for electrical cardioversion and if this intervention (regardless of rhythm conversion) could improve health-related quality of life in these patients.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common heart rhythm disorders worldwide. The estimated prevalence of AF in Europe is approximately 2% in the general population and increases with age, reaching 16-24% in individuals aged > 85 years. AF is significantly associated with an increased risk of heart failure, ischemic stroke, cognitive impairment, vascular dementia, and death. Aside from patient suffering, AF is a large economic burden for the healthcare system, where hospitalization is the major driver, accounting for 50-70% of the annual direct costs. Management of patients with AF is multifaceted. The main components include comorbidity and risk factor management (targeting hypertension, diabetes, heart failure), avoidance of stroke and thromboembolism, and reduction of symptoms through rate and rhythm control.

AF episodes may terminate spontaneously, and if they do so within seven days, they are classified as paroxysmal AF. Persistent AF is defined as AF episodes that are not self-terminating. Rhythm control, which involves restoring and maintaining sinus rhythm, is an important part of the management of patients with atrial fibrillation, where the main reason is to reduce symptoms of AF. One alternative treatment is electrical cardioversion (EC), which involves delivering low-energy shocks to the heart in a sedated patient to restore a normal sinus rhythm. A poorly tested alternative to EC in cardioversion is to physically increase the heart rate. In a small observational study, Gates et al. included 18 patients with AF scheduled for EC. The patients underwent a treadmill exercise test, and five (27.8%) converted to sinus rhythm during exercise. None of the patients who failed to convert to sinus rhythm with exercise did so spontaneously before electrical conversion 3 hours to 7 months later. Exercise tests are considered safe when contraindications are adhered to, termination criteria are observed, and appropriately trained personnel administer the tests.

Although EC is effective, it involves hospitalization, anesthesia, and the associated costs and risks. If exercise testing proves to be effective for converting AF to sinus rhythm, it could improve arrhythmia management by offering a non-invasive, cost-effective alternative that empowers patients to manage their condition through home-based programs. This approach not only would reduce hospital dependence and healthcare costs but also enhance cardiovascular fitness and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-75 years) with persistent AF
* planned for EC
* with at least 3 weeks of therapeutic oral anticoagulation before intervention

Exclusion Criteria:

* Unable to perform a symptom limited cycle exercise test
* Ischemic heart disease
* Heart failure
* Severe valvular disease
* Unable to speak and write Swedish language
* Unable to provide written, informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the pilot study - Recruitment rate | Day 1
  Number of patients asked to participate in the study
Feasibility of the pilot study - Consent rate | Day 1
  Number of patients giving written consent to participate in the study
Feasibility of the pilot study - Participant fidelity | From enrollment to the end of assessments, an average of 2 months
  Ability of participants to comply with the intervention protocol.
Feasibility of the pilot study - Study retention | Through study completion, an average of 6 months
  Participants dropout rates.
Feasibility of the pilot study - Adverse events | Through study completion, an average of 6 months
  Side effects and adverse events during the study

SECONDARY OUTCOMES:
AF conversion to sinus rhythm | Immediately after exercise or electrical conversion
  Rate of AF conversion to sinus rhythm immediately after intervention
Atrial fibrillation-related quality of life | At baseline and four weeks after intervention (exercise testing and/or electrical cardioversion)
  Atrial fibrillation-related quality of life, as measured by the AFEQT score.
Overall health-related quality of life | At baseline and four weeks after intervention (exercise testing and/or electrical cardioversion)
  Overall health-related quality of life, as measured by the EQ VAS (0-100) scale (from EQ5D-5L).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Research, Uppsala University, Västmanland County Hospital, Västerås, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Holmes DN, Piccini JP, Allen LA, Fonarow GC, Gersh BJ, Kowey PR, O'Brien EC, Reiffel JA, Naccarelli GV, Ezekowitz MD, Chan PS, Singer DE, Spertus JA, Peterson ED, Thomas L. Defining Clinically Important Difference in the Atrial Fibrillation Effect on Quality-of-Life Score. Circ Cardiovasc Qual Outcomes. 2019 May;12(5):e005358. doi: 10.1161/CIRCOUTCOMES.118.005358. PMID 31092022
- [Background] Gibbons L, Blair SN, Kohl HW, Cooper K. The safety of maximal exercise testing. Circulation. 1989 Oct;80(4):846-52. doi: 10.1161/01.cir.80.4.846. PMID 2791248
- [Background] Atterhog JH, Jonsson B, Samuelsson R. Exercise testing: a prospective study of complication rates. Am Heart J. 1979 Nov;98(5):572-9. doi: 10.1016/0002-8703(79)90282-5. PMID 495403
- [Background] Gates P, Al-Daher S, Ridley D, Black A. Could exercise be a new strategy to revert some patients with atrial fibrillation? Intern Med J. 2010 Jan;40(1):57-60. doi: 10.1111/j.1445-5994.2009.01940.x. PMID 19383061
- [Background] Van Gelder IC, Rienstra M, Bunting KV, Casado-Arroyo R, Caso V, Crijns HJGM, De Potter TJR, Dwight J, Guasti L, Hanke T, Jaarsma T, Lettino M, Lochen ML, Lumbers RT, Maesen B, Molgaard I, Rosano GMC, Sanders P, Schnabel RB, Suwalski P, Svennberg E, Tamargo J, Tica O, Traykov V, Tzeis S, Kotecha D; ESC Scientific Document Group. 2024 ESC Guidelines for the management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2024 Sep 29;45(36):3314-3414. doi: 10.1093/eurheartj/ehae176. No abstract available. PMID 39210723
- [Background] Wolowacz SE, Samuel M, Brennan VK, Jasso-Mosqueda JG, Van Gelder IC. The cost of illness of atrial fibrillation: a systematic review of the recent literature. Europace. 2011 Oct;13(10):1375-85. doi: 10.1093/europace/eur194. Epub 2011 Jul 14. PMID 21757483
- [Background] Dai H, Zhang Q, Much AA, Maor E, Segev A, Beinart R, Adawi S, Lu Y, Bragazzi NL, Wu J. Global, regional, and national prevalence, incidence, mortality, and risk factors for atrial fibrillation, 1990-2017: results from the Global Burden of Disease Study 2017. Eur Heart J Qual Care Clin Outcomes. 2021 Oct 28;7(6):574-582. doi: 10.1093/ehjqcco/qcaa061. PMID 32735316
- [Background] Mobley AR, Subramanian A, Champsi A, Wang X, Myles P, McGreavy P, Bunting KV, Shukla D, Nirantharakumar K, Kotecha D. Thromboembolic events and vascular dementia in patients with atrial fibrillation and low apparent stroke risk. Nat Med. 2024 Aug;30(8):2288-2294. doi: 10.1038/s41591-024-03049-9. Epub 2024 Jun 5. PMID 38839900
- [Background] Koh YH, Lew LZW, Franke KB, Elliott AD, Lau DH, Thiyagarajah A, Linz D, Arstall M, Tully PJ, Baune BT, Munawar DA, Mahajan R. Predictive role of atrial fibrillation in cognitive decline: a systematic review and meta-analysis of 2.8 million individuals. Europace. 2022 Sep 1;24(8):1229-1239. doi: 10.1093/europace/euac003. PMID 35061884
- [Background] Bassand JP, Accetta G, Al Mahmeed W, Corbalan R, Eikelboom J, Fitzmaurice DA, Fox KAA, Gao H, Goldhaber SZ, Goto S, Haas S, Kayani G, Pieper K, Turpie AGG, van Eickels M, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. Risk factors for death, stroke, and bleeding in 28,628 patients from the GARFIELD-AF registry: Rationale for comprehensive management of atrial fibrillation. PLoS One. 2018 Jan 25;13(1):e0191592. doi: 10.1371/journal.pone.0191592. eCollection 2018. PMID 29370229
- [Background] Ruddox V, Sandven I, Munkhaugen J, Skattebu J, Edvardsen T, Otterstad JE. Atrial fibrillation and the risk for myocardial infarction, all-cause mortality and heart failure: A systematic review and meta-analysis. Eur J Prev Cardiol. 2017 Sep;24(14):1555-1566. doi: 10.1177/2047487317715769. Epub 2017 Jun 15. PMID 28617620
- [Background] Odutayo A, Wong CX, Hsiao AJ, Hopewell S, Altman DG, Emdin CA. Atrial fibrillation and risks of cardiovascular disease, renal disease, and death: systematic review and meta-analysis. BMJ. 2016 Sep 6;354:i4482. doi: 10.1136/bmj.i4482. PMID 27599725
- [Background] Krijthe BP, Kunst A, Benjamin EJ, Lip GY, Franco OH, Hofman A, Witteman JC, Stricker BH, Heeringa J. Projections on the number of individuals with atrial fibrillation in the European Union, from 2000 to 2060. Eur Heart J. 2013 Sep;34(35):2746-51. doi: 10.1093/eurheartj/eht280. Epub 2013 Jul 30. PMID 23900699